CLINICAL TRIAL: NCT01531010
Title: Randomised Controlled Trial of Pressure-limited Ventilation Versus Volume-targeted Ventilation in Prematurely Born Infants
Brief Title: Pressure-limited Ventilation Versus Volume-targeted Ventilation in Preterm Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Anne Greenough, Professor of Neonatology and Clinical Respiratory Physiology, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/H0808/147-2
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Neonatal Respiratory Failure
Keywords: Neonate; Premature; Pressure limited ventilation; Volume ventilation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure-limited ventilation (Active Comparator)
  Interventions: Device: Ventilation protocol delivered by the SLE5000 ventilator
- Volume-targeted ventilation (Active Comparator)
  Interventions: Device: Ventilation protocol delivered by the SLE5000 ventilator

INTERVENTIONS:
Device: Ventilation protocol delivered by the SLE5000 ventilator — In pressure-limited ventilation arm, preferentially wean pressure till weaning criteria achieved, then wean rate.
  In volume-targeted ventilation arm, set target volume at 5ml/kg and wean rate. In both arms, aim to keep blood gases within normal limits.

SUMMARY:
Aims: There is increasing evidence that volume-targeted ventilation (VTV) holds benefits for preterm infants in comparison to pressure-limited ventilation. This study aims to compare pressure-limited to VTV in preterm infants.

Hypothesis: Volume-targeted will be associated with more rapid achievement of weaning criteria compared to pressure-limited ventilation

Primary outcome: Time taken to achieve pre-specified weaning criteria.

Methods: Ventilated infants less than 34 weeks gestational age at birth were recruited within the first 24 hours of life and randomly allocated to receive either pressure-limited or VTV. Adjustments to ventilator settings were made according to the trial protocol. Infants were deemed to have met failure criteria if they required HFOV, required peak pressures of more than 26 cm of water or developed pulmonary haemorrhage. Analysis will be by intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* <34 weeks gestation
* Within first 24 hours of life

Exclusion Criteria:

* Congenital diaphragmatic hernia
* Congenital heart disease
* Oesophageal atresia

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Time to achieve weaning criteria
  Peak inspiratory pressure (PIP) of 16 cm of water or less AND fraction of inspired oxygen of 0.4 or less for at least 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, London, United Kingdom